CLINICAL TRIAL: NCT00213018
Title: A Trial to Assess Expanded Safety, Acceptability and Preliminary Effectiveness of Carraguard™ (PC-515) in Preventing STI/HIV Transmission
Brief Title: Safety, Acceptability and Preliminary Effectiveness of Carraguard™ (PC-515) in Preventing HIV/STI Transmission
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Population Council (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); FHI 360 (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Medical Research Council, South Africa (Other); University of Cape Town (Other); University of Limpopo (Other); United States Agency for International Development (USAID) (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Population Council #210; R01AI045468-02 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2017-08-14 (Actual); Status verified 2017-08

CONDITIONS: HIV Infections; Chlamydia Trachomatis; Neisseria Gonorrhoeae; Trichomonas Vaginitis; Syphilis
Keywords: microbicides; HIV prevention; sexually transmitted infections; female-initiated protection; carrageenan; expanded safety trial; HIV Seronegativity; HIV
MeSH Terms: conditions — HIV Infections; Trichomonas Vaginitis; Syphilis; Sexually Transmitted Diseases

INTERVENTIONS:
Drug: Carraguard (PC-515)

SUMMARY:
The primary aims of the study were to assess the safety and acceptability of Carraguard ™ (PC-515) when applied vaginally at least three times weekly for 6-12 months. Secondary aims were to gather preliminary data on Carraguard's effectiveness in preventing male-to-female transmission of HIV.

The hypothesis was that Carraguard would cause little or no significant irritation, including lesions; that women would find Carraguard acceptable. The study was not powered to determine effectiveness, but based on safety, acceptability and feasibility parameters, the outcome of the Phase 2 trial would enable a decision whether or not to proceed to a Phase 3 efficacy trial.

DETAILED DESCRIPTION:
Carraguard™ (PC-515), the Population Council's lead candidate microbicide, was tested in a triple-masked, randomized, placebo-controlled trial fielded in two sites in South Africa. The primary aims of the study were to assess Carraguard's safety (toxicity) - including signs of irritation, such as itching or burning; changes in vaginal flora; and incidence of abnormal external genital, vaginal, and cervical findings - when applied vaginally for durations of 6-12 months, and to evaluate several dimensions of the acceptability of Carraguard and placebo products. Secondary aims were to investigate whether study participants using Carraguard had lower rates of HIV seroconversion or other sexually transmitted infections (including C. trachomatis, N. gonorrhoeae, T. vaginalis, and T. pallidum) than the placebo (methyl cellulose gel). In addition, when it began, this trial was the first to explore the feasibility of large-scale microbicides testing in a non-sex worker population. Last, the trial gauged women's reactions to using a non-contraceptive product (in vitro testing had shown that Carraguard has no contraceptive effect), as well as potential use-dynamics in communities where drying agents and other traditional vaginal products are used with high frequency.

ELIGIBILITY:
Inclusion Criteria:

* In good health as determined by medical history, physical examination and results of laboratory screening tests for RTIs
* Aged 18 years or older
* Resident in the area for at least one year and planning to stay for at least 12 months
* HIV-seronegative at screening
* Willing and able to comply with the study protocol (including being tested for HIV, learning the results, and undergoing clinical evaluations), and,
* Able to give informed consent

Exclusion Criteria:

* Pregnant or desire to become pregnant during the trial
* Delivered or aborted a pregnancy within the six weeks prior to screening
* History of surgery on external genitalia, vagina or cervix in the six weeks prior to screening
* Recent history of non-menstrual vaginal bleeding with intercourse
* Clinically detectable genital abnormality (including presence of warts, or a structural or congenital abnormality)
* Clinical suspicion of a RTI (defined as the presence of a genital ulcer visible to the naked eye, an abnormal vaginal discharge or purulent cervicitis, or untreated positive STI test result)
* Abnormal Pap smear
* History of sensitivity/allergy to latex
* Participating in another trial of a vaginal product
* Reported injection of recreational drugs

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 1999-10 (Actual); Study Completion 2002-01 (Actual)

PRIMARY OUTCOMES:
Safety (toxicity): Symptoms 14 days after enrollment and monthly thereafter (6-12 months); tests (monthly) to detect change in vaginal flora;
Compliance: collection of applicators and interview(monthly)
Acceptability: interview (quarterly)

SECONDARY OUTCOMES:
Preliminary effectiveness: Swabs taken to test for sexually transmitted infections - gonorrhea, chlamydia, trichomoniasis (monthly) and blood drawn for syphilis and HIV testing (Month 1 and quarterly thereafter).

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte E. Ellertson, MPA, Ph.D., Principal Investigator — Population Council
Locations (2):
- South Africa (2):
  - University of Cape Town, Department of Community Health, Cape Town
  - Medical University of Southern Africa, Soshanguve